CLINICAL TRIAL: NCT02952495
Title: Online Education to Inform the Elderly About Age-related Alcohol Risks: A Randomized Trial of Effectiveness and Costs
Brief Title: Online Education to Inform the Elderly About Age-related Alcohol Risks
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Arlene Fink Associates (Industry)
Collaborators: University of Southern California (Other)
Responsible Party: Principal Investigator, Arlene Fink, Principal Investigator, Arlene Fink Associates
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2R44AA022014-02 (NIH)
Record Dates: First submitted 2016-10-27; First posted 2016-11-02 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Alcohol Consumption; Drug-Food Interaction
Keywords: Alcohol Consumption; Older Adults
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Online alcohol educational class (Experimental): Participants will be asked to review an online alcohol education class. This is a web-based patient educational program designed to prevent hazardous and harmful drinking in older adults.
  Interventions: Behavioral: Online alcohol educational class
- No intervention (No Intervention): Participants will NOT Participate in the online alcohol education class.

INTERVENTIONS:
Behavioral: Online alcohol educational class — Participants will be asked to review an online alcohol education class. This is a web-based patient educational program designed to prevent hazardous and harmful drinking in older adults. The project's specific objectives are to 1) provide reliable information on the extent to which "A Toast to Health in Later Life!" reduces alcohol-related risks and problems among older patients who drink and 2) evaluate the extent to which these reductions are associated with increases in health-related quality of life, patient knowledge and self-efficacy and decreases in the use of health services and the costs of care.
  Arms: Online alcohol educational class

SUMMARY:
This proposed Phase 2 The Small Business Innovation Research study is a randomized trial of the effectiveness of "A Toast to Health in Later Life!" a web-based patient educational program designed to prevent hazardous and harmful drinking in older adults. The project's specific objectives are to

1. provide reliable information on the extent to which "A Toast to Health in Later Life!" reduces alcohol-related risks and problems among older patients who drink and
2. evaluate the extent to which these reductions are associated with increases in health-related quality of life, patient knowledge and self-efficacy and decreases in the use of health services and the costs of care.

DETAILED DESCRIPTION:
This proposed Phase 2 The Small Business Innovation Research study is a randomized trial of the effectiveness of "A Toast to Health in Later Life!" a web-based patient educational program designed to prevent hazardous and harmful drinking in older adults. The project's specific objectives are to 1) provide reliable information on the extent to which "A Toast to Health in Later Life!" reduces alcohol-related risks and problems among older patients who drink and 2) evaluate the extent to which these reductions are associated with increases in health-related quality of life, patient knowledge and self-efficacy and decreases in the use of health services and the costs of care. The proposal is being submitted in response to the The National Institute on Alcohol Abuse and Alcoholism's interest in the "development and evaluation of educational materials designed to intervene with the elderly around specific age-related risks for alcohol problems" and to the National Institute of Health's highest priority areas in health economics research because it aims to measure the actual or potential impact of a specific intervention "on healthcare utilization and health outcomes." The study will take place with 600 patients who currently drink and receive their care at a large community-based medical center in in L.A. County that serves a stable and diverse population. Older people can experience alcohol's unfavorable health effects even at relatively low consumption levels because of age-related physiological changes and drinking's potentially adverse interactions with chronic illness, increased medication-use and diminishing functional status. About 14.5% of older adults drink in excess of the The National Institute on Alcohol Abuse and Alcoholism's recommended limits. Excessive alcohol consumption is responsible for an average of 88,000 deaths and 2.5 million years of potential life lost each year in the U.S. and cost the 50 States a median of $2.9 billion in 2006. Most of the costs are due to binge drinking. According to The Centers for Disease Control and Prevention, older adults binge-drink more frequently than their younger counterparts, and drinking too much contributes to over 54 different injuries and diseases (including car crashes and violence). Further, the chance of getting sick and dying from alcohol problems increases significantly for those who binge drink more often. When health and drinking patterns are accounted for, about half of all older drinkers may be at risk for experiencing alcohol-related harm even if they drink within recommended limits. Considering that about 10,000 people will turn 65 every day for the next decade, and that the proportion of older adults will increase to more than 20% of the U.S. population by 2030, the number of older people with alcohol-related risks will increase even if drinking prevalence remains constant. Despite this, many physicians fail to discuss drinking with older patients, partly because they do not have the time and training to do so and partly because the available education focuses on younger drinkers. To complicate matters, observational evidence suggests that in some older adults, moderate consumption may have beneficial effects on cardiovascular functioning and mortality. "A Toast to Health in Later Life!" covers the spectrum of drinking and its benefits and risks. If effective and cost-effective, the product has the potential to achieve important clinical and societal benefits.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older
* have had one or more drinks containing alcohol in the past 3 months
* have an active email account
* have access to high-speed Internet
* are able and willing to spend about 30 minutes on three separate occasions to complete an online alcohol use class and answer questions in English

Exclusion Criteria:

* Non alcohol drinkers (having no drinks containing alcohol in the past 3 months)

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-09; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Alcohol Risk Score Baseline | Alcohol Risk Score at Baseline
  Health and drinking patterns are accounted at baseline
Alcohol Risk Score 6 months | Change from Baseline Alcohol Risk Score at 6 months
  Health and drinking patterns are accounted at 6 months

SECONDARY OUTCOMES:
Costs and cost effectiveness | Six months
  Costs of achieving changes in drinking patterns and risks

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Fink, Principal Investigator — Arlene Fink Associates
Locations (1):
- Arlene Fink Associates, Pacific Palisades, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fink A, Kwan L, Osterweil D, Van Draanen J, Cooke A, Beck JC. Assessing the Usability of Web-Based Alcohol Education for Older Adults: A Feasibility Study. JMIR Res Protoc. 2016 Feb 1;5(1):e11. doi: 10.2196/resprot.4545. PMID 26832213
- See also: Fink A, Kwan L, Osterweil D, Van Draanen J, Cooke A, Beck JC. Assessing the Usability of Web-Based Alcohol Education for Older Adults: A Feasibility Study. JMIR Res Protoc. 2016 Feb 1;5(1):e11. doi: 10.2196/resprot.4545. — http://www.researchprotocols.org/2016/1/e11/